CLINICAL TRIAL: NCT03051607
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Tolerability of Tozadenant as Adjunctive Therapy in Levodopa-Treated Patients With Parkinson's Disease Experiencing End of Dose "Wearing-Off"
Brief Title: Safety and Tolerability of Tozadenant as Adjunctive Therapy in Levodopa-Treated Patients With Parkinson's Disease.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New Safety Information
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOZ-CL06
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Motor Fluctuations; Off time; On time; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — tozadenant

STUDY DESIGN:
Intervention Model Description: Eligible patients will begin dosing with tozadenant at a dose of 120 mg twice daily. At Week 2 or thereafter, the investigator may adjust the patient's IMP dose as clinically indicated; doses of 60 mg BID and 120 mg BID will be permitted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tozadenant (Experimental): 120 mg twice daily. At Week 2 or thereafter doses of 60 mg BID and 120 mg BID will be permitted.
  Interventions: Drug: Tozadenant

INTERVENTIONS:
Drug: Tozadenant — 1 Year Open Label, 120 mg BID tozadenant, with dose modification to 60 mg BID tozadenant permitted.
  Other Names: SYN115

SUMMARY:
Phase 3, international, multicenter, open-label 12 month safety study.

DETAILED DESCRIPTION:
Each patient will participate for up to 52 weeks, which includes a Screening Period, followed by a Baseline Visit and open-label treatment for 1 year with a safety Follow-up 4 weeks after the last treatment.

* Screening Period: up to 6 weeks.
* Open-Label Treatment Period: 52 weeks (1 year)
* Post-Treatment Safety Follow Up: 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands study requirements and has given his/her written informed consent on an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved consent form.
* Parkinson's disease diagnosis consistent with UK Parkinson's Disease Society Brain Bank Diagnostic criteria
* Minimum of 3 years since diagnosis.
* Meet Hoehn and Yahr PD stage
* Good response to levodopa
* Stable regimen of anti-PD medications
* Patients must have been taking a levodopa-containing anti-PD medication continuously for at least the previous 12 months
* Patient has documented a minimum amount of Off time.
* If of childbearing potential (male and female) must use an acceptable method of contraception

Exclusion Criteria:

* Previous tozadenant study participation
* Current or recent participation in another study.
* Secondary or atypical parkinsonism
* Neurosurgical intervention for PD (except DBS if electrode placement has been performed over 12 months prior to screening)
* Patient is taking apomorphine, budipine, istradefylline, tolcapone, or DUOPA™/Duodopa®
* Treatment with excluded medications
* Untreated or uncontrolled hyperthyroidism or hypothyroidism
* Clinically significant out-of-range laboratory
* MMSE out of range
* Current episode of major depression (stable treatment for depression is permitted).
* Recent suicide attempt or suicidal ideation type 4 or type 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Women lactating or pregnant
* Hypersensitivity to any components of tozadenant or excipients
* Abnormal findings on the physical or neurological examination, or medical history that would make the patient unsuitable for the study
* History of hepatitis or cholangitis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kenney, MD, Study Director — Acorda Therapeutics
Locations (33):
- United States (29):
  - Barrow Neurology Clinics, St. Joseph's Hospital and Medical Center, Dignity Health, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - USC, Keck School of Medicine, Los Angeles, California
  - SC3 Research Group, Pasadena, California
  - JEM Research Institute, Atlantis, Florida
  - Aventura Neurologic Associates, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Infinity Clinical Research, Sunrise, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Unity Point Health, Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Department of Neurology, Lexington, Kentucky
  - Henry Ford West Bloomfield Hospital, Bloomfield Hills, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - The Robert and John M. Bendheim Parkinson and Movement Disorders Center, New York, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Movement Disorders Clinic of Oklahoma, Tulsa, Oklahoma
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Department of Neurology, Charlottesville, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Premier Clinical Research, Spokane, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
  - University of Wisconsin - Madison, Madison, Wisconsin
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada
- United Kingdom (3):
  - The Walton Centre NHS Foundation Trust, Neuroscience Research Center, Liverpool, England
  - Newcastle University Clinical Ageing Research Unit (CARU), Newcastle upon Tyne, England
  - The Queen Elizabeth University Hospital Department of Neurology, Glasgow, Scottland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The disposition of study patients. A total of 66 patients were enrolled in 27 study centers across 6 countries: USA, United Kingdom, Italy, Canada, Spain and Hungary, and were included in the Safety Set (SS) as well as the Full Analysis Set (FAS).
Period: Overall Study
Arm/Group | Tozadenant
Started | 66
Completed | 0
Not Completed | 66
Not completed — Adverse Event | 66

BASELINE CHARACTERISTICS:
Population: Planned patient enrollment numbers were not achieved as this study and the tozadenant development program were terminated early, based on an unexpected emerging safety signal. A total of 60 out of 66 enrolled patients completed up to Week 2, 44 completed Week 4, 22 completed Week 12, and 4 completed Week 24.
Arm/Group | Tozadenant
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 61
  Black or African American | 1
  Asian | 3
  American Indian or Alaska Native | 1
  Hispanic or Latino | 6
  Not Hispanic or Latino | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51
  United Kingdom | 6
  Canada | 1
  Spain | 1
  Hungary | 1
  Italy | 6
Weight at Screening [Mean (Standard Deviation); unit: kg] | 80.4 (17.18)

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety and Tolerability of Tozadenant in Levodopa-treated PD Patients Experiencing Motor Fluctuations.
Description: The primary objective of this study was to evaluate the safety and tolerability of tozadenant in levodopa-treated Parkinson's Disease (PD) patients experiencing motor fluctuations, based on assessment of treatment-emergent adverse events (TEAEs), vital signs, electrocardiograms (ECGs), and clinical laboratory tests. A total of 66 patients were enrolled in 27 study centers across 6 countries: USA, United Kingdom, Italy, Canada, Spain and Hungary, and were included in the Safety Set (SS).
Time Frame: Up to 28 Weeks including safety follow-up visit.
Population: Safety evaluation was based on Safety Set which included all 66 patients enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozadenant
Number analyzed (Participants) | 66
Participants
  Subjects with at least one treatment-emergent AE | 46
  Subjects with at least one related TEAE | 33
  Subjects discontinuing study drug due to an AE | 7
  Subjects with at least one SAE | 5
  Subjects with at least one life-threatening SAE | 5
  Subjects with AE leading to death | 2

2. Secondary Outcome: To Evaluate the Effects of Tozadenant on the Occurrences of Daytime Drowsiness by Using the Epworth Sleepiness Scale.
Description: The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a short questionnaire. Minimum range is 0 - Maximum range is 24. A score within the range 0-9 is considered to be normal while a score within the range of 10-24 would indicate that medical help should be solicited.
Time Frame: Up to 28 Weeks including safety follow-up visit.
Population: Planned patient enrollment numbers were not achieved as this study and the tozadenant development program were terminated early, based on an unexpected emerging safety signal. No patient completed the 52 Week study treatment period prior to Sponsor termination of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tozadenant
Number analyzed (Participants) | 66
score on a scale
  Baseline | 7.9 (5.32)
  Week 2: number analyzed (Participants) | 59
  Week 2 | 7.4 (5.29)
  Week 6: number analyzed (Participants) | 44
  Week 6 | 8.5 (4.72)
  Week 12: number analyzed (Participants) | 22
  Week 12 | 10.0 (3.53)
  Week 24: number analyzed (Participants) | 4
  Week 24 | 12.0 (4.08)
  Early Termination: number analyzed (Participants) | 61
  Early Termination | 7.9 (5.08)
  Safety Follow-up: number analyzed (Participants) | 56
  Safety Follow-up | 7.3 (4.95)

3. Secondary Outcome: To Evaluate the Effects of Tozadenant on the Number of Participants With Suicidal Ideation or Behavior Using the Columbia-Suicide Severity Scale (C-SSRS) Summarized by Visit.
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is a standardized suicidality rating system. The interview measures presence of suicidality and consists of 4 categories: suicidal ideation, intensity of ideation, suicidal behavior, and actual/potential lethality.
  Suicidal Ideation - A series of 1 -5 questions with 5 types of ideation of increasing severity. Score of Yes = 1, No= 0. A positive answer to question 4 (active suicidal ideation with some intent to act) or 5 (active suicidal ideation with specific plan and intent) indicates that the individual has some intent to act on suicidal thoughts and will need further evaluation.
  Suicidal Behavior - Different types of suicidal behavior are scored (Yes=1, No=0) and identify the occurrence of actual, interrupted, or aborted attempts; preparatory behaviors; and suicide. The total number of each type of suicidal behavior show the density of suicide, (more behaviors represent a higher degree of risk).
Time Frame: Up to 28 Weeks including safety follow-up visit.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tozadenant
Number analyzed (Participants) | 66
Participants
  Screening - Lifetime: Actual attempts | 2
  Screening - Lifetime: Interrupted attempts | 2
  Screening - Lifetime: Aborted attempts | 3
  Screening - Past 5 years: Actual attempts | 2
  Screening - Past 5 years: Interrupted attempts | 2
  Screening - Past 5 years: Aborted attempts | 2
  Screening - Past 6 months: Actual attempts | 2
  Screening - Past 6 months: Interrupted attempts | 2
  Screening - Past 6 months: Aborted attempts | 2
  Baseline - Since last visit: Actual attempts | 3
  Baseline - Since last visit: Interrupted attempts | 2
  Baseline - Since last visit: Aborted attempts | 3
  Week 2 - Since last visit: Actual attempts | 3
  Week 2 - Since last visit: Interrupted attempts | 3
  Week 2 - Since last visit: Aborted attempts | 3
  Week 6 - Since last visit: Actual attempts | 1
  Week 6 - Since last visit: Interrupted attempts | 1
  Week 6 - Since last visit: Aborted attempts | 1
  Week 12 - Since last visit: Actual attempts | 1
  Week 12 - Since last visit: Interrupted attempts | 1
  Week 12 - Since last visit: Aborted attempts | 1
  Week 24 - Since last visit: Actual attempts | 1
  Week 24 - Since last visit: Interrupted attempts | 1
  Week 24 - Since last visit: Aborted attempts | 1
  Early Termination: Actual attempts | 10
  Early Termination: Interrupted attempts | 10
  Early Termination: Aborted attempts | 10
  Safety Follow-up: Actual attempts | 8
  Safety Follow-up: Interrupted attempts | 8
  Safety Follow-up: Aborted attempts | 11

4. Secondary Outcome: To Evaluate the Effects of Tozadenant on the Number of Participants With Occurrence of Impulsive Behavior - Modified Minnesota Impulse Disorder Interview (mMIDI)
Description: The Minnesota Impulsive Disorders Interview (MIDI) 8 is a global instrument that includes questions for compulsive gambling, buying, and sexual behavior (as well as other disorders not reported to occur in PD).
  The mMIDI consists of 5 modules: compulsive buying, compulsive gambling, compulsive eating, hypersexuality and punding.
  Positive Answer: Any answer other than "no" on any question is considered a "yes"/positive answer.
  Negative Module: A module is considered negative if the patient's answer to a gateway (initial) question is "no" or if a patient answers "yes" to a gateway question and "no" to all of the remaining answers after the gateway question in that module.
  Positive Module: A module is considered positive if a patient gives a positive answer (No = 0, rarely = 1, occasionally = 2, frequently = 3) to any question after the gateway (initial) question in one or more of the 5 modules.
Time Frame: Up to 28 Weeks including safety follow-up visit.
Population: Planned patient enrollment numbers were not achieved as this study and the tozadenant development program were terminated early, based on an unexpected emerging safety signal. No patient completed the 52 Week study treatment period prior to Sponsor termination of the study. .
Measure: Count of Participants; unit: Participants
Arm/Group | Tozadenant
Number analyzed (Participants) | 66
Participants
  Buying Disorder - Screening: Negative | 66
  Buying Disorder - Screening: Positive | 0
  Buying Disorder - Week 2: number analyzed (Participants) | 60
  Buying Disorder - Week 2: Negative | 59
  Buying Disorder - Week 2: Positive | 1
  Buying Disorder - Week 6: number analyzed (Participants) | 44
  Buying Disorder - Week 6: Negative | 43
  Buying Disorder - Week 6: Positive | 1
  Buying Disorder - Week 12: number analyzed (Participants) | 22
  Buying Disorder - Week 12: Negative | 22
  Buying Disorder - Week 12: Positive | 0
  Buying Disorder - Week 24: number analyzed (Participants) | 4
  Buying Disorder - Week 24: Negative | 4
  Buying Disorder - Week 24: Positive | 0
  Buying Disorder - Early Termination: number analyzed (Participants) | 62
  Buying Disorder - Early Termination: Negative | 60
  Buying Disorder - Early Termination: Positive | 2
  Buying Disorder - Safety Follow-up: number analyzed (Participants) | 57
  Buying Disorder - Safety Follow-up: Negative | 56
  Buying Disorder - Safety Follow-up: Positive | 1
  Compulsive Gambling - Screening: Negative | 65
  Compulsive Gambling - Screening: Positive | 1
  Compulsive Gambling - Week 2: number analyzed (Participants) | 60
  Compulsive Gambling - Week 2: Negative | 59
  Compulsive Gambling - Week 2: Positive | 1
  Compulsive Gambling - Week 6: number analyzed (Participants) | 44
  Compulsive Gambling - Week 6: Negative | 44
  Compulsive Gambling - Week 6: Positive | 0
  Compulsive Gambling - Week 12: number analyzed (Participants) | 22
  Compulsive Gambling - Week 12: Negative | 22
  Compulsive Gambling - Week 12: Positive | 0
  Compulsive Gambling - Week 24: number analyzed (Participants) | 4
  Compulsive Gambling - Week 24: Negative | 4
  Compulsive Gambling - Week 24: Positive | 0
  Compulsive Gambling - Early Termination: number analyzed (Participants) | 62
  Compulsive Gambling - Early Termination: Negative | 61
  Compulsive Gambling - Early Termination: Positive | 1
  Compulsive Gambling - Safety Follow-up: number analyzed (Participants) | 57
  Compulsive Gambling - Safety Follow-up: Negative | 56
  Compulsive Gambling - Safety Follow-up: Positive | 1
  Compulsive Sexual Behavior - Screening: Negative | 66
  Compulsive Sexual Behavior - Screening: Positive | 0
  Compulsive Sexual Behavior - Week 2: number analyzed (Participants) | 60
  Compulsive Sexual Behavior - Week 2: Negative | 60
  Compulsive Sexual Behavior - Week 2: Positive | 0
  Compulsive Sexual Behavior - Week 6: number analyzed (Participants) | 44
  Compulsive Sexual Behavior - Week 6: Negative | 44
  Compulsive Sexual Behavior - Week 6: Positive | 0
  Compulsive Sexual Behavior - Week 12: number analyzed (Participants) | 22
  Compulsive Sexual Behavior - Week 12: Negative | 22
  Compulsive Sexual Behavior - Week 12: Positive | 0
  Compulsive Sexual Behavior - Week 24: number analyzed (Participants) | 4
  Compulsive Sexual Behavior - Week 24: Negative | 4
  Compulsive Sexual Behavior - Week 24: Positive | 0
  Compulsive Sexual Behavior - Early Termination: number analyzed (Participants) | 62
  Compulsive Sexual Behavior - Early Termination: Negative | 60
  Compulsive Sexual Behavior - Early Termination: Positive | 2
  Compulsive Sexual Behavior - Safety Follow-up: number analyzed (Participants) | 57
  Compulsive Sexual Behavior - Safety Follow-up: Negative | 56
  Compulsive Sexual Behavior - Safety Follow-up: Positive | 1
  Compulsive Eating Module - Screening: Negative | 66
  Compulsive Eating Module - Screening: Positive | 0
  Compulsive Eating Module - Week 2: number analyzed (Participants) | 60
  Compulsive Eating Module - Week 2: Negative | 60
  Compulsive Eating Module - Week 2: Positive | 0
  Compulsive Eating Module - Week 6: number analyzed (Participants) | 44
  Compulsive Eating Module - Week 6: Negative | 43
  Compulsive Eating Module - Week 6: Positive | 1
  Compulsive Eating Module - Week 12: number analyzed (Participants) | 22
  Compulsive Eating Module - Week 12: Negative | 22
  Compulsive Eating Module - Week 12: Positive | 0
  Compulsive Eating Module - Week 24: number analyzed (Participants) | 4
  Compulsive Eating Module - Week 24: Negative | 4
  Compulsive Eating Module - Week 24: Positive | 0
  Compulsive Eating Module - Early Termination: number analyzed (Participants) | 62
  Compulsive Eating Module - Early Termination: Negative | 61
  Compulsive Eating Module - Early Termination: Positive | 1
  Compulsive Eating Module - Safety Follow-up: number analyzed (Participants) | 57
  Compulsive Eating Module - Safety Follow-up: Negative | 57
  Compulsive Eating Module - Safety Follow-up: Positive | 0
  Punding Behavior - Screening: Negative | 66
  Punding Behavior - Screening: Positive | 0
  Punding Behavior - Week 2: number analyzed (Participants) | 60
  Punding Behavior - Week 2: Negative | 60
  Punding Behavior - Week 2: Positive | 0
  Punding Behavior - Week 6: number analyzed (Participants) | 44
  Punding Behavior - Week 6: Negative | 44
  Punding Behavior - Week 6: Positive | 0
  Punding Behavior - Week 12: number analyzed (Participants) | 22
  Punding Behavior - Week 12: Negative | 22
  Punding Behavior - Week 12: Positive | 0
  Punding Behavior - Week 24: number analyzed (Participants) | 4
  Punding Behavior - Week 24: Negative | 4
  Punding Behavior - Week 24: Positive | 0
  Punding Behavior - Early Termination: number analyzed (Participants) | 62
  Punding Behavior - Early Termination: Negative | 62
  Punding Behavior - Early Termination: Positive | 0
  Punding Behavior - Safety Follow-up: number analyzed (Participants) | 57
  Punding Behavior - Safety Follow-up: Negative | 57
  Punding Behavior - Safety Follow-up: Positive | 0

ADVERSE EVENTS:
Time Frame: This study and the tozadenant development program were terminated early, based on an unexpected emerging safety signal. Due to Sponsor termination of the study, Adverse Events were collected up to Week 24.
Arm/Group | Tozadenant
All-Cause Mortality (participants affected / at risk) | 2/66
Serious Adverse Events (participants affected / at risk) | 5/66
Other Adverse Events (participants affected / at risk) | 46/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tozadenant (N=66)
Agranulocytosis (Blood and lymphatic system disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tozadenant (N=66)
Dyskinesia (Nervous system disorders) | 17
Fall (Injury, poisoning and procedural complications) | 7
Nausea (Gastrointestinal disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 4
Diarrhea (Gastrointestinal disorders) | 3
Hallucination (Psychiatric disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Parkinson's Disease (Nervous system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Agranulocytosis (Blood and lymphatic system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Blood pressure increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Drug administration error (Injury, poisoning and procedural complications) | 2
Headache (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
Tremor (Nervous system disorders) | 2
Urinary tract infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT03051607/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03051607/SAP_001.pdf